CLINICAL TRIAL: NCT06856525
Title: Dissolved Phase Hyperpolarized Xenon-129 MRI: a Novel Biomarker to Quantify Pulmonary Pathology in Young Healthy E-cigarette Users
Brief Title: Dissolved Phase HXe-129 MRI: a Novel Biomarker to Quantify Pulmonary Pathology in Young Healthy E-cigarette Users
Acronym: ECIG
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Y. Michael Shim, MD (Other)
Collaborators: Duke University (Other); George Mason University (Other)
Responsible Party: Sponsor-Investigator, Y. Michael Shim, MD, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 230348
Record Dates: First submitted 2024-11-15; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Electronic Cigarette Related Lung Damage
Keywords: hyperpolarized xenon-129 MRI; cardiopulmonary stress test; lung damage; vaping; healthy young adult
MeSH Terms: conditions — Vaping | interventions — Exercise Test; Respiratory Function Tests

STUDY DESIGN:
Intervention Model Description: 40 Participants who are healthy with less than 6 months of smoking history and electronic cigarette users with more than 6 months of electronic cigarette usage. Subjects will be recruited and consented at the University of Virginia and Duke University.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Participants (Other): Young, healthy subjects without any lung disease or other inflammatory diseases.
  Interventions: Drug: Hyperpolarized Xe129; Diagnostic Test: Cardiopulmonary Stress Test; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Chest CT
- eCig user (Experimental): Young, otherwise healthy subjects who have used electronic cigarettes for at least 6 months past year.
  Interventions: Drug: Hyperpolarized Xe129; Diagnostic Test: Cardiopulmonary Stress Test; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Chest CT

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Determine the impact of e-cigarette use on pulmonary gas exchange capacity in interstitial tissues and capillaries using hyperpolarized xenon-129 MRI.
Diagnostic Test: Cardiopulmonary Stress Test — Exercise stress test to evaluate cardiac and pulmonary fitness.
  Other Names: CPET
Diagnostic Test: Pulmonary Function Test — Standard clinic pulmonary function test to evaluate lung function
  Other Names: PFT
Diagnostic Test: Chest CT — Clinical standard chest computer tomography to evaluate any lung tissue scars or air movement.

SUMMARY:
A two-center, longitudinal assessment of 40 electronic cigarette users and 40 healthy controls at the initial visit and a follow-up visit 12 months later. This study will determine the impact of electronic cigarette use on pulmonary gas exchange capacity and then corroborate the Hyperpolarized Xenon MRI (HXeMRI) results with the cardiopulmonary stress test at the initial visit and a follow-up visit 12 months later.

DETAILED DESCRIPTION:
Electronic cigarettes have been commercialized as a "less harmful" alternative to traditional cigarettes. Electronic cigarettes generate vapor from ingredients containing well-known toxic materials such as carbonyls, tobacco-specific N-nitrosamines, and heavy metals. Nonhuman studies show that Electronic cigarettes cause pulmonary epithelial, endothelial, and vascular dysfunction. Electronic cigarette use has also been associated with cardiac and pulmonary diseases, including severe respiratory failure. Our preliminary studies suggest that we can detect subtle early changes in healthy young e-cigarette users by hyperpolarized xenon-129 MR imaging. We anticipate the following results from the three primary analyses. First, there will be significantly impaired gas exchange in electronic cigarette users compared to healthy controls at the initial and follow-up visits. Second, gas exchange impairment in electronic cigarette users will increase after an additional 12 months of electronic cigarette use. Further, as a secondary analysis, we speculate that because electronic cigarette users exhaust their cardiopulmonary reserve at rest, they will have reduced physical fitness detectable by the 6-minute walk and Cardio-pulmonary exercise tests.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 35 years old.
2. At their baseline health
3. Ability to understand a written informed consent form and comply with the requirements of the study.
4. Exclusive long-term, recent, and greater than six months continuous e-cigarette use with greater than three days a week frequency.
5. Users of "closed-container" and "pre-packaged" electronic cigarette juices that must contain nicotine.
6. At baseline, normal spirometry with or without bronchodilator, plethysmograph lung volume, carbon monoxide diffusion capacity, and 6-minute walk by ATS/ERS with Global Lung Initiative Reference.

   -

Exclusion Criteria:

1. History of any other lung disease
2. History of brain diseases including stroke and dementia, end-stage liver disease, coronary artery disease, renal failure
3. Acute infection of any kind previous 6 weeks
4. Pregnancy or a possibility of pregnancy
5. Anemia
6. Inability to undergo PFT, CPET, or MR imaging (usual clinical standard criteria for MRI)
7. Prior cigarette smoking of greater than one pack-year within six months before enrolling in the study.
8. Using a non-closed container, custom-made electronic cigarette juice, or inability for the study team to access "closed-container" and "pre-packaged" electronic cigarette juice for chemical analysis
9. Significant history of smoking other substances in the past year.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between e-cig user vs. healthy participants at baseline and 12 month later | baseline and 12 month follow-up
  Hyperpolarized MRI (ventilation defect, RBC/Gas, Membrane/Gas, and RBC/membrane numbers) capillaries using HXeMRI, and corroborate the HXeMRI signatures with the CPET for 40 young adults with ecigarette use at an initial visit (V1) and a follow-up visit 12-months later (V2).
Acute effects of e-cig in e-cig users before and after using one usual dose at baseline and 12 months follow-up | baseline and 12 months follow-up
  Cardiopulmonary stress test maximum oxygen uptake
Acute effects of e-cig in e-cig users before and after using one usual dose at baseline and 12 months follow-up | Baseline and 12 months follow up
  Pulmonary Function Test with 6 minute walk test

SECONDARY OUTCOMES:
Acute Effects of eCig use at baseline and 12 months follow-up | baseline and 12 months follow-up
  blood levels of 32 chemical toxins

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
As a part of publications.